CLINICAL TRIAL: NCT01733459
Title: The Role of DLBS3233 in the Management of Polycystic Ovary Syndrome (PCOS)
Brief Title: Efficacy and Safety of DLBS3233 in Subjects With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS3233-0811
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: PCOS, DLBS3233, metformin,oral anti-hyperglycemic agent
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — DLBS3233

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment I (Experimental): 1 DLBS3233 capsule 100 mg (once daily) and 1 placebo caplet of Metformin XR (twice daily)
  Interventions: Drug: DLBS3233; Drug: Placebo caplet of Metformin XR
- Treatment II (Active Comparator): 1 Metformin XR caplet 750 mg (twice daily) and 1 placebo capsule of DLBS3233 (once daily)
  Interventions: Drug: Metformin XR; Drug: Placebo capsule of DLBS3233

INTERVENTIONS:
Drug: DLBS3233 — 1 DLBS3233 capsule 100 mg once daily for 6 months
  Other Names: Inlacin
  Arms: Treatment I
Drug: Metformin XR — 1 Metformin XR caplet 750 mg twice daily for 6 months
  Other Names: Glumin XR
  Arms: Treatment II
Drug: Placebo caplet of Metformin XR — 1 placebo caplet of Metformin XR twice daily for 6 months
  Other Names: Placebo caplet of Glumin XR
  Arms: Treatment I
Drug: Placebo capsule of DLBS3233 — 1 placebo capsule of DLBS3233 once daily for 6 months
  Other Names: Placebo capsule of Inlacin
  Arms: Treatment II

SUMMARY:
This is a 2-arm, randomized, double-blind, double-dummy, and controlled clinical study, with 6 months of treatment to evaluate the clinical and metabolic efficacy of DLBS3233 in improving reproductive parameters and to evaluate the safety of DLBS3233 in women with polycystic ovary syndrome compared with metformin, as an active control.

DETAILED DESCRIPTION:
There will be 2 groups of treatment; each group will consist of 62 subjects with the treatment regimens :

* Treatment I : 1 capsule of DLBS3233 100 mg (once daily) and 1 placebo caplet of Metformin XR (twice daily)
* Treatment II : 1 caplet of Metformin XR 750 mg (twice daily) and 1 placebo capsule of DLBS3233 (once daily) for 6 months of treatment.

Clinical examination to evaluate the efficacy of the investigational drug will be performed at baseline and every interval of 1 month.

Laboratory examinations to evaluate the metabolic efficacy parameters and ultrasonography (USG) examination will be performed at baseline, Month 3rd, and end of study (Month 6th). In addition to that, USG will also be performed about 2 weeks after Month 3rd (Month 3.5th) and after Month 5th (Month 5.5th).

Laboratory examinations to evaluate the reproductive efficacy parameters (reproductive hormone levels) and safety, at baseline and Month 6th (end of study).

General counseling on lifestyle modification will be provided to the subjects by the assigned Nutritionist. All study subjects should follow a lifestyle modification. Evaluation on subjects' performance on lifestyle modification will be conducted every follow-up visit by Investigator, but particularly at baseline, Month 3rd, and end of study (Month 6th) by the Nutritionist.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects in reproductive age (i.e. 18-40 years)
* Subject with a diagnosis of polycystic ovary syndrome confirmed by two of the Rotterdam Criteria
* Subject with insulin resistance defined by: HOMA-IR of > 2.00

Exclusion Criteria:

* Pregnant and lactating women
* Subjects known to have Cushing's syndrome, late onset of congenital adrenal hyperplasia, androgen-secreting tumors, uncontrolled thyroid disease, hyperprolactinemia
* Known to have current medical condition, which, is judged by the Investigator could jeopardize subject's health or interfere with the study evaluation, such as diabetes mellitus, uncontrolled hypertension, other cardiovascular diseases, acute or chronic infections, and any known malignancies
* Impaired renal function (serum creatinine level > 1.5 ULN)
* Impaired liver function (serum ALT level ≥ 2.5 ULN)
* Medically-assisted weight loss with medications or surgical procedures
* Currently having laparoscopic ovarian diathermy (LOD)
* Currently under treatment with in vitro fertilization (IVF) techniques
* Have been regularly taking any medications which affect insulin sensitivity as well as reproductive function (i.e. ovulation, menstrual cycle), within ≤ 3 months prior to screening
* Participating in other clinical trial within 30 days prior to screening

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2013-03; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
HOMA-IR reduction | 6 months
  HOMA-IR reduction from baseline to Month 6th (end of study)

SECONDARY OUTCOMES:
Reduction of S/A ratio | 3 and 6 months
  Reduction (indicating improvement) of S/A ratio (i.e. ratio of mean stromal echogenicity to mean echogenicity of entire ovary) from baseline to Month 3rd and Month 6th (end of study)
Reduction of free testosterone level (calculated) | 6 months
  Reduction of free testosterone level (calculated) from baseline to Month 6th (end of study)
Change of luteinizing hormone (LH) level | 6 months
  Change of luteinizing hormone (LH) level from baseline to Month 6th (end of study)
Change of luteinizing hormone (LH) / follicle stimulating hormone (FSH) ratio | 6 months
  Change of luteinizing hormone (LH) / follicle stimulating hormone (FSH) ratio from baseline to Month 6th (end of study)
Change of Ferriman-Gallwey Score | 3 and 6 months
  Change of Ferriman-Gallwey Score from baseline to Month 3rd and Month 6th (end of study)
Improvement of glucose tolerance | 3 and 6 months
  Improvement of glucose tolerance (reduction of FPG and 2-hour PPPG) from baseline to Month 3rd and Month 6th (end of study)
Fasting insulin level reduction | 3 and 6 months
  Fasting insulin level reduction from baseline to Month 3rd and Month 6th (end of study)
HOMA-IR reduction | 3 months
  HOMA-IR reduction from baseline to Month 3rd
Lipid profile improvement | 3 and 6 months
  Lipid profile improvement (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides level) from baseline to Month 3rd and Month 6th (end of study)
Liver function | 6 months
  Liver function (serum AST, ALT, alkaline phosphatase, γ-glutamyl transferase) from baseline to Month 6th (end of study)
Renal function | 6 months
  Renal function (serum creatinine, BUN) from baseline to Month 6th (end of study)
Number of adverse events and subjects with events | During 6 months
  Adverse events as well as number of events and subjects experiencing the events will be observed and evaluated throughout study period (6 months) and until all adverse events have been recovered or stabilized

CONTACTS AND LOCATIONS:
Overall Officials: Andon Hestiantoro, dr., SpOG(K), Principal Investigator — Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia; Wiryawan Permadi, Dr., dr., SpOG(K), Principal Investigator — Department of Obstetrics and Gynecology, Faculty of Medicine, University of Padjadjaran, Hasan Sadikin Hospital, Bandung, Indonesia
Locations (2):
- Indonesia (2):
  - Department of Obstetrics and Gynecology, Faculty of Medicine, University of Padjadjaran, Hasan Sadikin Hospital, Bandung, West Java
  - Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta

REFERENCES:
- [Derived] Hestiantoro A, Permadi W, Tjandrawinata RR, Wiweko B, Ritonga MA, Ferrina AI, Sumapraja K, Muharam R, Djuwantono T. The Efficacy and Safety of DLBS3233, A Combined Bioactive Fraction of Cinnamomum burmanii and Lagerstroemia speciosa Plants on The Endocrine-Metabolic Profile of Women with Polycystic Ovary Syndrome: A Randomized Clinical Trial. Int J Fertil Steril. 2024 Jul 13;18(Suppl 1):35-47. doi: 10.22074/ijfs.2023.551350.1283. PMID 39033369